CLINICAL TRIAL: NCT05528887
Title: Safety and Efficacy Study of Chimeric Antigen Receptor T (CAR-T) Cells in the Treatment of Relapsed/Refractory Hematological Malignancies
Brief Title: Study of CAR-T Cell Therapy in the Treatment of Relapsed/Refractory Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated People's Hospital of Ningbo University (Other Government)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-037
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Relapsed/Refractory Hematological Malignancies; Lymphoma; Myeloma; Leukemia
Keywords: CD19 CAR-T; BCMA CAR-T; CD7 CAR-T; CD123 CAR-T
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Neoplasms, Plasma Cell; Leukemia | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous CAR-T cells (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CAR-T cells. CAR-T cells targeted CD19/BCMA/CD123/CD7 are autologous genetically modified T cells.
  Interventions: Biological: Autologous CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Autologous CAR-T cells — D0: CAR-T cells will be infused intravenously.
Drug: Fludarabine — D-5 to D-3: Fludarabine (30 mg/m^2/day) will be administered intravenously for 3 days.
  Other Names: Fludara
Drug: Cyclophosphamide — D-5 to D-3: Cyclophosphamide (500 mg/m^2/day) will be administered intravenously for 3 days.
  Other Names: Cytoxan

SUMMARY:
The primary purpose of this study is to determine the safety and efficacy of novel autologous CAR-T cells in patients with relapsed/refractory hematological malignancies.

DETAILED DESCRIPTION:
CAR-T cells targeted CD19 have demonstrated unprecedented successes. Besides CD19, many other molecules such as CD123, BCMA, and CD7 may be potential in developing the corresponding CAR-T cells to treat patients with hematopoietic and lymphoid malignancies. UTC Therapeutics Inc. have developed an efficient platform for constructing CAR-T cells that can remodel of tumor microenvironment and enhance the anti-tumor immune response and persistence of CAR-T cells. In this study, all eligible subjects will receive a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by investigational treatment, CAR-T cells. Safety and efficacy of the CAR-T cells will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of hematological malignancies (such as lymphoma, myeloma, leukemia) refractory to, or relapsing after standard therapy.
2. Positive expression of specific antigens.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0~2.
4. Adequate organ functions:

   * Serum bilirubin ≤ 35 μmol/L;
   * Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 2;
   * Serum creatinine (Cr) ≤ 2 × upper limit of normal (ULN);
   * Brain natriuretic peptide (BNP)<80 pg/mL.
5. Subjects must be able to understand the protocol and be willing to enroll the study, sign the informed consent, and be able to comply with the study and follow-up procedures.

Exclusion Criteria:

1. History of allergy to any of the drugs involved in the protocol.
2. History of cardiac diseases:

   * Left ventricular ejection fraction (LVEF) < 50%;
   * Class III or IV heart failure as defined by the New York Heart Association (NYHA).
3. History of another malignancy tumor.
4. Active hepatitis C (HCV), hepatitis B (HBV), human immunodeficiency virus (HIV), or syphilis infection.
5. Patients with any contraindications to allogeneic hematopoietic stem cell transplantation.
6. Uncontrolled fungal, bacterial, viral, or other infection.
7. Female subjects who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
TEAEs | 4 weeks
  Incidence and severity of Treatment Emergent Adverse Event.
TRAEs | 4 weeks
  Incidence and severity of Treatment Related Adverse Events.
AESIs | 4 weeks
  Incidence and severity of AEs of Special Interest.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (PR+CR) | 12 months
  The proportion of patients with complete response(CR) or partial response(PR)
Progression-Free Survival (PFS) | 12 months
  PFS was defined as the time from CAR-T infusion to the date of disease progression or death from any cause.
  Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Overall survival (OS) | 12 months
  OS was defined as the time from CAR-T infusion to the date of death. Participants who did not die by the analysis data cutoff date were censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Lu, Principal Investigator — The Affiliated People's Hospital of Ningbo University
Locations (1):
- The Affiliated People's Hospital of Ningbo University, Ningbo, Zhejiang, China